CLINICAL TRIAL: NCT00649480
Title: Single-Dose Fed Bioequivalence Study of Balsalazide Disodium Capsules (750 mg; Mylan) and Colazal® Capsules (750 mg; Salix) in Healthy Volunteers
Brief Title: Fed Study of Balsalazide Disodium Capsules 750 mg and Colazal® Capsules 750 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BALS-06128
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — balsalazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): BALSALAZIDE DISODIUM CAPSULES, 750 MG
  Interventions: Drug: BALSALAZIDE DISODIUM CAPSULES, 750 MG
- 2 (Active Comparator): COLAZAL® Capsules 750 mg
  Interventions: Drug: COLAZAL® Capsules 750 mg

INTERVENTIONS:
Drug: BALSALAZIDE DISODIUM CAPSULES, 750 MG — 3x750mg, single dose fed
  Arms: 1
Drug: COLAZAL® Capsules 750 mg — 3x750mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan balsalazide disodium 750 mg capsules to Salix Colazal® 750 mg capsules following a single, oral 2250 mg (3 x 750 mg) dose administration under fed conditions.

DETAILED DESCRIPTION:
This open-label, single dose, randomized, two-period, two-treatment, two-sequence, crossover study was conducted to investigate the bioequivalence of two formulations of balsalazide disodium 750 mg capsules under non-fasting conditions. The study was conducted with 60 (60 completing) healthy adults in accordance with Protocol No. BALS-06128 (Version 22 December 2006). In each study period, a single, oral 2250 mg dose (3 x 750 mg capsules) was administered to all subjects following an overnight fast of at least 10 hours. The test formulation was Mylan Pharmaceuticals Inc.'s Balsalazide Disodium Capsules, 750 mg and the reference formulation was Colazal® 750 mg capsules (manufactured for Salix Pharmaceuticals, Inc.). The subjects received the test product in one study period and the reference product in the other study period. Drug administration occurred according to the dosing randomization schedule (see Appendix 16.1.7). There was a 7-day washout interval between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 years and older
* Sex: Male and/or non-pregnant, non-lactating female
* Women of childbearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 21 days prior to the start of the study and on the evening prior to each dose administration An additional serum (β-HCG) pregnancy test was performed upon completion of the study
* Women of childbearing potential were required to practice abstinence or use an acceptable form of contraception throughout the duration of the study No hormonal contraceptives or hormonal replacement therapies were permitted in this study Acceptable forms of contraception included the following
* intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period or
* barrier methods containing or used in conjunction with a spermicidal agent or surgical sterilization
* Women were not considered of childbearing potential if one of the following was reported and documented on the medical history
* postmenopausal with an absence of menses for at least one (1) year or
* bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months or
* total hysterectomy
* During the course of the study from study screen until study exit including the washout period all men and women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive method
* Weight:At least(132 lbs) for men and(106 lbs) for women with all subjects having a Body Mass Index less than or equal to 30 but greater than or equal to 19
* All subjects were judged normal and healthy during a pre-study medical evaluation (physical examination laboratory evaluation Hepatitis B and Hepatitis C tests HIV test 12-lead ECG and urine drug screen including amphetamine barbiturates benzodiazepines cannabinoid cocaine opiates phencyclidine and methadone) performed within 21 days of the initial dose of study medication

Exclusion Criteria:

* Institutionalized subjects were not used
* Use of any tobacco-containing products within 1 year of the start of the study
* Ingestion of any alcoholic caffeine or xanthine containing food or beverage within the 48 hours prior to the initial dose of study medication
* Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication
* Any recent significant change in dietary or exercise habits
* A positive test for any drug included in the urine drug screen
* History of drug and or alcohol abuse
* Use of any prescription or over-the-counter medications within the 14 days prior to the initial dose of study medication
* Use of any hormonal contraceptives or hormone replacement therapy within 3 months prior to study medication dosing
* Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication
* History of any significant cardiovascular hepatic renal pulmonary hematologic gastrointestinal endocrine immunologic dermatologic or neurologic disease
* Acute illness at the time of either the pre-study medical evaluation or dosing
* A positive HIV hepatitis B or hepatitis C test
* Abnormal and clinically significant laboratory test results
* Clinically significant deviation from the Guide to Clinically Relevant
* Abnormal and clinically relevant ECG tracing
* Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication
* Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication
* Allergy or hypersensitivity to balsalazide disodium salicylates or other related products
* History of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption
* Consumption of grapefruit or grapefruit containing products within 7 days of drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Copa, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html